CLINICAL TRIAL: NCT06563219
Title: Comparative Analysis of Traditional Clinical Scores and Combined Grading Systems in Predicting 28-Day Mortality in Non-Traumatic Subarachnoid Hemorrhage
Brief Title: Predicting 28-Day Mortality in Subarachnoid Hemorrhage
Acronym: SAHstdy
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Az, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: 38-2024
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Subarachnoid Hemorrhage; Aneurysmal; Non-traumatic; Glasgow coma scale; World federation of neurological surgeons scale; modified Fisher scale; VASOGRADE scale; Ogilvy-Carter scale; 28-day mortality
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Glasgow Coma Scale; Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Survivors were defined as patients who were still alive after 28 days of admission to the emergency department.
  Interventions: Other: Glasgow coma scale; Other: Hunt-Hess scale; Other: World Federation of Neurological Surgeons (WFNS) scale; Other: modified Fisher scale; Other: VASOGRADE scale; Other: Ogilvy and Carter scale
- Non-survivors: Non-survivors had passed away within 28 days of admission to the emergency department.
  Interventions: Other: Glasgow coma scale; Other: Hunt-Hess scale; Other: World Federation of Neurological Surgeons (WFNS) scale; Other: modified Fisher scale; Other: VASOGRADE scale; Other: Ogilvy and Carter scale

INTERVENTIONS:
Other: Glasgow coma scale — The levels of response in the components of the Glasgow Coma Scale are 'scored' from 1, for no response, up to normal values of 4 (Eye-opening response) 5 ( Verbal response) and 6 (Motor response) The total Coma Score thus has values between three and 15, three being the worst and 15 being the highest.
Other: Hunt-Hess scale — The Hunt-Hess scale was used to assess SAH severity according to the clinical presentation and the visible neurological deficits. The Grades run from 1 to 5:
  * Grade 1: Asymptomatic or minimal headache, slight neck stiffness.
  * Grade 2: Moderate to severe headache, and neck stiffness, but no neurological deficit except cranial nerve palsy.
  * Grade 3: Drowsiness, confusion, or a mild focal deficit.
  * Grade 4: Stupor, moderate to severe hemiparesis, early decerebrate rigidity, and vegetative disturbance.
  * Grade 5: Deep coma, decerebrate rigidity, and a moribund appearance.
Other: World Federation of Neurological Surgeons (WFNS) scale — The World Federation of Neurological Surgeons (WFNS) scale, introduced in 1988, is used to evaluate the clinical severity of patients with SAH. This scale is derived from the GCS score and considers the presence of motor deficits:
  * Grade 1: GCS score of 15, no motor deficit
  * Grade 2: GCS score of 13 to 14, no motor deficit
  * Grade 3: GCS score of 13 to 14, with motor deficit
  * Grade 4: GCS score of 7 to 12, with or without motor deficit
  * Grade 5: GCS score of 3 to 6, with or without motor deficit
Other: modified Fisher scale — The modified Fisher scale was used to evaluate SAH severity by reference to the extent of hemorrhage as revealed by CT of the brain. Four grades are depending on the degree of bleeding observed:
  * Grade 0: No hemorrhage apparent in CT.
  * Grade 1: Minimal hemorrhage without intraventricular hemorrhage (IVH).
  * Grade 2: Thin or diffusely thin (<1mm) hemorrhage with bilateral IVH.
  * Grade 3: Thick (> 1 mm) hemorrhage without bilateral IVH.
  * Grade 4: Thick (> 1 mm) hemorrhage with bilateral IVH.
Other: VASOGRADE scale — The VASOGRADE scale was established to estimate the risk of delayed cerebral ischemia following SAH. This scale is based on the WFNS and the modified Fisher scales at admission. There are three categories:
  * Green: WFNS score of 1 or 2 and modified Fisher scale of 1 or 2.
  * Yellow: WFNS score of 1 or 3 and modified Fisher scale of 3 or 4.
  * Red: WFNS score of 4 or 5 and any modified Fisher scale score.
Other: Ogilvy and Carter scale — The Ogilvy and Carter scale is a grading system used to predict the outcomes of surgical treatment in patients with SAH due to a ruptured aneurysm. The scale considers multiple factors, including age, Hunt and Hess grade, Fisher grade, and aneurysm size, with a score assigned to each of these variables:
  * Age greater than 50
  * Hunt and Hess grade of 4 to 5
  * Fisher grade scores of 3 to 4
  * Aneurysm size >10 mm
  * An additional point is added for a giant posterior circulation aneurysm (≥25 mm)

SUMMARY:
The investigators investigated the predictive ability of clinical and radiological scores, including the Glasgow coma scale (GCS), Hunt-Hess, World Federation of Neurological Surgeons (WFNS), and modified Fisher scales, as well as combined clinical scores such as the VASOGRADE and Ogilvy-Carter rating scales, for 28-day mortality in patients presenting to the emergency department (ED) with non-traumatic subarachnoid hemorrhage (SAH). Specifically, we tested the hypothesis that combined clinical scores are more reliable and superior to non-combined clinical and radiological scores in predicting 28-day mortality in non-traumatic SAH.

DETAILED DESCRIPTION:
Patients were divided into survivors and non-survivors, with surviving patients further categorized as either mobile or immobile based on the Glasgow outcome scale. Accordingly, patients who were dependent on daily support or in a coma were classified as immobile, whereas patients who had returned to normal life or were independent in their daily activities were classified as mobile. The demographic (age and sex), comorbidities (hypertension, diabetes mellitus [DM] and/or coronary artery disease [CAD]), vital signs (systolic blood pressure, heart rate, respiratory rate, and peripheral capillary oxygen saturation [sPO2]), and clinical assessment tools (GCS, Hunt Hess, WFNS, modified Fisher, VASOGRADE, and Ogilvy-Carter rating scales) on admission were compared between the groups to identify factors associated with 28-day mortality and neurological survival. Independent predictors of mortality were determined by multivariate logistic regression analysis of variables (demographic characteristics, clinical characteristics, and trauma scores) that differed significantly between survivors and non-survivors. An area under the curve (AUC) analysis was then conducted to identify which trauma score is the most reliable and superior predictor of mortality.

ELIGIBILITY:
Inclusion Criteria:

* patients (aged ≥ 18 years) who presented to the emergency department with non-traumatic Subarachnoid Hemorrhage between September 2020 and September 2023

Exclusion Criteria:

* patients younger than 18 years
* patients with missing information
* patients with traumatic SAH
* patients with subdural or epidural hemorrhage
* patients with concurrent ischemic stroke

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This multicenter, retrospective, observational cohort study enrolled 451 consecutive adult patients (aged ≥ 18 years) who presented to the emergency departments of the six major and highest-volume tertiary hospitals in Istanbul with non-traumatic Subarachnoid Hemorrhage between September 2020 and September 2023. Data were collected by searching for I60.9 International Classification of Disease (ICD) codes in the hospital's automation systems and archives.
Sampling Method: Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Predictive ability of Glasgow coma scale for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of Glasgow coma scale in determining 28-day mortality.
Predictive ability of Hunt-Hess scale for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of Hunt-Hess scale in determining 28-day mortality.
Predictive ability of World Federation of Neurological Surgeons (WFNS) scale for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of World Federation of Neurological Surgeons (WFNS) scale in determining 28-day mortality.
Predictive ability of modified Fisher scale for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of modified Fisher scale in determining 28-day mortality.
Predictive ability of VASOGRADE scale for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of VASOGRADE scale in determining 28-day mortality.
Predictive ability of Ogilvy-Carter rating scale for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of Ogilvy-Carter rating scale in determining 28-day mortality.

SECONDARY OUTCOMES:
Predictive ability of Glasgow coma scale for neurological survival | From admission to 28 days
  The investigators assessed the predictive ability of Glasgow coma scale in determining neurological survival
Predictive ability of Hunt-Hess scale for neurological survival | From admission to 28 days
  The investigators assessed the predictive ability of Hunt-Hess scale in determining neurological survival
Predictive ability of World Federation of Neurological Surgeons (WFNS) scale for neurological survival | From admission to 28 days
  The investigators assessed the predictive ability of World Federation of Neurological Surgeons (WFNS) scale in determining neurological survival
Predictive ability of modified Fisher scale for neurological survival | From admission to 28 days
  The investigators assessed the predictive ability of modified Fisher scale in determining neurological survival
Predictive ability of VASOGRADE scale for neurological survival | From admission to 28 days
  The investigators assessed the predictive ability of VASOGRADE scale in determining neurological survival
Predictive ability of Ogilvy-Carter rating scale for neurological survival | From admission to 28 days
  The investigators assessed the predictive ability of Ogilvy-Carter rating scale in determining neurological survival

CONTACTS AND LOCATIONS:
Overall Officials: Adem Az, M.D., Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Stored in non-publicly available Available on request

REFERENCES:
- [Result] Sharma D. Perioperative Management of Aneurysmal Subarachnoid Hemorrhage. Anesthesiology. 2020 Dec 1;133(6):1283-1305. doi: 10.1097/ALN.0000000000003558. PMID 32986813
- [Result] Hijdra A, van Gijn J, Nagelkerke NJ, Vermeulen M, van Crevel H. Prediction of delayed cerebral ischemia, rebleeding, and outcome after aneurysmal subarachnoid hemorrhage. Stroke. 1988 Oct;19(10):1250-6. doi: 10.1161/01.str.19.10.1250. PMID 3176085
- [Result] Rosen DS, Macdonald RL. Subarachnoid hemorrhage grading scales: a systematic review. Neurocrit Care. 2005;2(2):110-8. doi: 10.1385/NCC:2:2:110. PMID 16159052
- [Result] Ogilvy CS, Carter BS. A proposed comprehensive grading system to predict outcome for surgical management of intracranial aneurysms. Neurosurgery. 1998 May;42(5):959-68; discussion 968-70. doi: 10.1097/00006123-199805000-00001. PMID 9588539
- [Result] Takagi K, Tamura A, Nakagomi T, Nakayama H, Gotoh O, Kawai K, Taneda M, Yasui N, Hadeishi H, Sano K. How should a subarachnoid hemorrhage grading scale be determined? A combinatorial approach based solely on the Glasgow Coma Scale. J Neurosurg. 1999 Apr;90(4):680-7. doi: 10.3171/jns.1999.90.4.0680. PMID 10193613
- [Result] Dengler NF, Sommerfeld J, Diesing D, Vajkoczy P, Wolf S. Prediction of cerebral infarction and patient outcome in aneurysmal subarachnoid hemorrhage: comparison of new and established radiographic, clinical and combined scores. Eur J Neurol. 2018 Jan;25(1):111-119. doi: 10.1111/ene.13471. Epub 2017 Nov 2. PMID 28940973